CLINICAL TRIAL: NCT04237857
Title: Long Term Incidence and Effect of Gastroesophageal Reflux Disease After Laparoscopic Sleeve Gastrectomy in Chinese Population
Brief Title: Long Term Incidence and Effect of de Novo GERD After Laparoscopic Sleeve Gastrectomy in Chinese Population
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Cheung Yau Fung, Associate Consultant, Chinese University of Hong Kong
Other Study IDs: CRE-2019.362
Record Dates: First submitted 2020-01-17; First posted 2020-01-23 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Gastroesophageal Reflux
Keywords: Sleeve gastrectomy; Gastroesophageal reflux; Chinese
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LSG: Chinese patients who received laparoscopic sleeve gastrectomy at Prince of Wales Hospital, The Chinese University of Hong Kong for more than 36 months
  Interventions: Procedure: Laparoscopic sleeve gastrectomy

INTERVENTIONS:
Procedure: Laparoscopic sleeve gastrectomy — Laparoscopic sleeve gastrectomy

SUMMARY:
To evaluate the long-term incidence and effects of gastroesophageal reflux disease in the Chinese population after laparoscopic sleeve gastrectomy.

DETAILED DESCRIPTION:
Laparoscopic sleeve gastrectomy (SG) has gained popularity as a primary bariatric procedure in the past decade. According to the International Federation for the Surgery of Obesity and Metabolic Disorders (IFSO), 43.6% of all bariatric procedures performed worldwide were SG between 2013 and 2017. Long term data of SG have shown that the procedure is able to achieve adequate weight loss and metabolic outcomes compared with other bariatric procedures. Furthermore, it has gained popularity due to its relatively simpler procedure, shorter operative time, avoidance of intestinal anatomy rearrangement, anastomosis, risk of internal hernia, and lower risk of malnutrition.

One major drawback to SG is potential development of gastrointestinal reflux disease (GERD). According to the Montreal Classification, GERD is defined as heartburn and regurgitation because of reflux contents of the stomach into the esophagus, causing symptoms that interferes with physical activity, disturbs sleep and reduce productivity at work . It has been shown to significant impact on patients' post-operative quality of life negatively . Currently there are discrepancy in the medical literature, while some studies found worsening of GERD or development of GERD (de novo GERD) after SG, some found improvement of GERD post-operatively. From a recent meta-analysis by Yeung et al comprising 10, 718 patients with follow-up period from 3 to 132 months, 19% of patients experienced worsening of GERD while 23% developed de novo GERD after SG.

Furthermore, long term complications of GERD include the development of erosive esophagitis, Barret's esophagus and even esophageal adenocarcinoma. From the same meta-analysis, the long-term prevalence (>24 months) of erosive esophagitis and Barret's esophagus were 28% and 8% respectively. There have also been isolated case reports of development of esophageal adenocarcinoma after SG. From the investigators' literature review, four cases were reported. Two of the cases had no pre-operative endoscopy, one case had pre-operative diagnosis of Barret's esophagus. The other case developed esophageal adenocarcinoma despite normal pre-operative endoscopy 5 years after SG.

The epidemiology of GERD is different in Western countries and in Asian countries. Although the incidence of GERD has increased in the past decades, the prevalence of GERD was 5.2-8.5% base on symptoms. Prevalence of Barret's esophagus remained rare at 0.06-0.85%. In patents who have received SG, Tai et al showed that the prevalence of GERD increased from 12.1 to 47% based on Reflux Disease Questionnaire at one year after SG. The prevalence of erosive esophagitis also increased from 16.7 to 66.7%. based on upper gastrointestinal endoscopy findings at one year. In the long run, the prevalence of de novo GERD was 17-45% based on symptoms and proton pump inhibitors use from the case series by Pok et al. and Chang et al. with a follow-up period up to 7 years and 10 years respectively.

From the current Asian literature, data on long term incidence of GERD after SG based on objective assessment tools and endoscopy findings was lacking. There is also no adequate data on the long-term occurrence of erosive esophagitis and Barret's esophagus after SG, which would have important significance in pre-operative counselling.

The objective of the study is to evaluate the long-term incidence and effects of gastroesophageal reflux disease in the Chinese population after laparoscopic sleeve gastrectomy.

ELIGIBILITY:
Inclusion Criteria:

* Chinese patients who received laparoscopic sleeve gastrectomy at Prince of Wales Hospital, The Chinese University of Hong Kong
* SG has been performed more than 36 months
* Patient received preoperative OGD and GI symptom assessment with C-GIQLI questionnaire
* Willing and able to consent to the study

Exclusion Criteria:

* Revisional surgery
* Concomitant surgeries (except hiatal repair/ cholecystectomy)
* Mentally incompetent patients or patients less than 18 years old
* Pregnant patients
* Inmates
* Unable/unwilling to consent to the study
* Unable/unwilling to undergo follow-up assessments

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Chinese patients who received laparoscopic sleeve gastrectomy at Prince of Wales Hospital, The Chinese University of Hong Kong for more than 36 months
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of de novo GERD | >36 months after surgery
  Incidence of long term de novo gastroesophageal reflux disease after laparoscopic sleeve gastrectomy, as defined by: Patients who did not have pre-operative GERD; AND patients who scored ≥12 in the Chinese GERDQ questionnaire at ≥36 months after SG; and/or patients who scored ≤5 out of 8 marks in questions 26 (acid reflux) and 34 (heart burn), at ≥36 months after SG; and/or patients who had erosive esophagitis or Barret's esophagus at upper gastrointestinal endoscopy at ≥36 months after SG; and/or patients who required regular anti-reflux medications at ≥36 months after SG

SECONDARY OUTCOMES:
Changes in severity of GERD | >36 months after surgery
  Changes in severity of GERD after SG in patients who had pre-operative GERD, defined by increase in anti-reflux medications usage and/or increase in severity of erosive esophagitis or Barret's esophagus at ≥36 months after SG
Proportion of asymptomatic patients with endoscopic evidence of de novo GERD | >36 months after surgery
  Proportion of patients who have endoscopic evidence of de novo GERD (erosive esophagitis or Barret's esophagus) but had no symptoms of de novo GERD
Difference in quality of life in patient with or without de novo GERD | >36 months after surgery
  Difference in quality of life as measured by C-GIQLI questionnaire between patients who have de novo GERD and patients who do not at ≥36 months after operation

CONTACTS AND LOCATIONS:
Overall Officials: Yau Fung Cheung, FRCSEd(Gen), Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yeung KTD, Penney N, Ashrafian L, Darzi A, Ashrafian H. Does Sleeve Gastrectomy Expose the Distal Esophagus to Severe Reflux?: A Systematic Review and Meta-analysis. Ann Surg. 2020 Feb;271(2):257-265. doi: 10.1097/SLA.0000000000003275. PMID 30921053
- [Background] Peterli R, Wolnerhanssen BK, Peters T, Vetter D, Kroll D, Borbely Y, Schultes B, Beglinger C, Drewe J, Schiesser M, Nett P, Bueter M. Effect of Laparoscopic Sleeve Gastrectomy vs Laparoscopic Roux-en-Y Gastric Bypass on Weight Loss in Patients With Morbid Obesity: The SM-BOSS Randomized Clinical Trial. JAMA. 2018 Jan 16;319(3):255-265. doi: 10.1001/jama.2017.20897. PMID 29340679
- [Background] Salminen P, Helmio M, Ovaska J, Juuti A, Leivonen M, Peromaa-Haavisto P, Hurme S, Soinio M, Nuutila P, Victorzon M. Effect of Laparoscopic Sleeve Gastrectomy vs Laparoscopic Roux-en-Y Gastric Bypass on Weight Loss at 5 Years Among Patients With Morbid Obesity: The SLEEVEPASS Randomized Clinical Trial. JAMA. 2018 Jan 16;319(3):241-254. doi: 10.1001/jama.2017.20313. PMID 29340676
- [Background] Vakil N, van Zanten SV, Kahrilas P, Dent J, Jones R; Global Consensus Group. The Montreal definition and classification of gastroesophageal reflux disease: a global evidence-based consensus. Am J Gastroenterol. 2006 Aug;101(8):1900-20; quiz 1943. doi: 10.1111/j.1572-0241.2006.00630.x. PMID 16928254
- [Background] Felsenreich DM, Prager G, Kefurt R, Eilenberg M, Jedamzik J, Beckerhinn P, Bichler C, Sperker C, Krebs M, Langer FB. Quality of Life 10 Years after Sleeve Gastrectomy: A Multicenter Study. Obes Facts. 2019;12(2):157-166. doi: 10.1159/000496296. Epub 2019 Mar 15. PMID 30879011
- [Background] Popescu AL, Ionita-Radu F, Jinga M, Gavrila AI, Savulescu FA, Fierbinteanu-Braticevici C. Laparoscopic sleeve gastrectomy and gastroesophageal reflux. Rom J Intern Med. 2018 Dec 1;56(4):227-232. doi: 10.2478/rjim-2018-0019. PMID 30521478
- [Background] Braghetto I, Csendes A. Prevalence of Barrett's Esophagus in Bariatric Patients Undergoing Sleeve Gastrectomy. Obes Surg. 2016 Apr;26(4):710-4. doi: 10.1007/s11695-015-1574-1. PMID 25855575
- [Background] Felsenreich DM, Kefurt R, Schermann M, Beckerhinn P, Kristo I, Krebs M, Prager G, Langer FB. Reflux, Sleeve Dilation, and Barrett's Esophagus after Laparoscopic Sleeve Gastrectomy: Long-Term Follow-Up. Obes Surg. 2017 Dec;27(12):3092-3101. doi: 10.1007/s11695-017-2748-9. PMID 28593484
- [Background] El Khoury L, Benvenga R, Romero R, Cohen R, Roussel J, Catheline JM. Esophageal adenocarcinoma in Barrett's esophagus after sleeve gastrectomy: Case report and literature review. Int J Surg Case Rep. 2018;52:132-136. doi: 10.1016/j.ijscr.2018.10.015. Epub 2018 Oct 12. PMID 30343262
- [Background] Wright FG, Duro A, Medici JR, Lenzi S, Beskow AF, Cavadas D. Esophageal adenocarcinoma five years after laparoscopic sleeve gastrectomy. A case report. Int J Surg Case Rep. 2017;32:47-50. doi: 10.1016/j.ijscr.2017.01.054. Epub 2017 Feb 11. PMID 28235650
- [Background] Jung HK. Epidemiology of gastroesophageal reflux disease in Asia: a systematic review. J Neurogastroenterol Motil. 2011 Jan;17(1):14-27. doi: 10.5056/jnm.2011.17.1.14. Epub 2011 Jan 26. PMID 21369488
- [Background] Tai CM, Huang CK, Lee YC, Chang CY, Lee CT, Lin JT. Increase in gastroesophageal reflux disease symptoms and erosive esophagitis 1 year after laparoscopic sleeve gastrectomy among obese adults. Surg Endosc. 2013 Apr;27(4):1260-6. doi: 10.1007/s00464-012-2593-9. Epub 2012 Dec 12. PMID 23232995
- [Background] Pok EH, Lee WJ, Ser KH, Chen JC, Chen SC, Tsou JJ, Chin KF. Laparoscopic sleeve gastrectomy in Asia: Long term outcome and revisional surgery. Asian J Surg. 2016 Jan;39(1):21-8. doi: 10.1016/j.asjsur.2015.03.006. Epub 2015 May 8. PMID 25964106
- [Background] Chang DM, Lee WJ, Chen JC, Ser KH, Tsai PL, Lee YC. Thirteen-Year Experience of Laparoscopic Sleeve Gastrectomy: Surgical Risk, Weight Loss, and Revision Procedures. Obes Surg. 2018 Oct;28(10):2991-2997. doi: 10.1007/s11695-018-3344-3. PMID 29931481
- [Background] Kasama K, Mui W, Lee WJ, Lakdawala M, Naitoh T, Seki Y, Sasaki A, Wakabayashi G, Sasaki I, Kawamura I, Kow L, Frydenberg H, Chen A, Narwaria M, Chowbey P. IFSO-APC consensus statements 2011. Obes Surg. 2012 May;22(5):677-84. doi: 10.1007/s11695-012-0610-7. PMID 22367008
- [Background] Yeung SM, Shiu AT, Martin CR, Chu KM. Translation and validation of the Chinese version of the Gastrointestinal Quality of Life Index in patients with gastric tumor. J Psychosom Res. 2006 Oct;61(4):469-77. doi: 10.1016/j.jpsychores.2006.03.049. PMID 17011354
- [Background] Wong WM, Lam KF, Lai KC, Hui WM, Hu WH, Lam CL, Wong NY, Xia HH, Huang JQ, Chan AO, Lam SK, Wong BC. A validated symptoms questionnaire (Chinese GERDQ) for the diagnosis of gastro-oesophageal reflux disease in the Chinese population. Aliment Pharmacol Ther. 2003 Jun 1;17(11):1407-13. doi: 10.1046/j.1365-2036.2003.01576.x. PMID 12786635